CLINICAL TRIAL: NCT01057199
Title: Critical Role of MicroRNA-34a and MicroRNA-194 in Acute Myeloid Leukemia With CEBPA Mutations
Brief Title: Studying Biomarkers in Cell Samples From Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B13; COG-AAML10B13 (Other: Children's Oncology Group); CDR0000664229 (Other: Clinical Trials.gov); NCI-2011-02207 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia; childhood acute myeloid leukemia/other myeloid malignancies
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Gene Expression Profiling; Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — cell samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: protein expression analysis
Other: fluorescence activated cell sorting
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at biomarkers in cell samples from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the significance of regulation of microRNA-34a and microRNA-194 by C/EBPα during granulopoiesis in patients with acute myeloid leukemia with CEBPA mutations.
* To determine whether overexpression of micro RNA-34a and microRNA-194 in myeloid progenitors with C/EBPα mutations leads to granulocytic differentiation.
* To examine how microRNA-34a and microRNA-194 downregulate E2F3 during granulopoiesis.
* To determine the role of microRNA-34a and microRNA-194 in myeloid cell proliferation.

OUTLINE: Cryopreserved cell samples are collected for laboratory analysis, including mutation analysis, gene expression analysis, RNA analysis, and fluorescence-activated cell sorting (FACS) analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia with CEBPA mutations

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of acute myeloid leukemia with CEBPA mutations
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Significance of regulation of microRNA-34a and microRNA-194 by C/EBPα during granulopoiesis
Relationship between overexpression of microRNA-34a and microRNA-194 in myeloid progenitors with C/EBPα mutations and granulocytic differentiation
Downregulation of E2F3 by microRNA-34a and microRNA-194 during granulopoiesis
Role of microRNA-34a and microRNA-194 in myeloid cell proliferation

CONTACTS AND LOCATIONS:
Overall Officials: Soheil Meshinchi, MD, Principal Investigator — Fred Hutchinson Cancer Center